CLINICAL TRIAL: NCT06321913
Title: Phase II Study to Evaluate the Safety, Tolerability and Efficacy of IBI343 Combined With Sintilimab in Subjects With Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of IBI343 in Subjects With Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Yanqiao Zhang, chief physician, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI343Y002
Record Dates: First submitted 2024-02-23; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI343 (Experimental)
  Interventions: Drug: IBI343 combined with IBI308

INTERVENTIONS:
Drug: IBI343 combined with IBI308 — IBI343 Specifications: 100 mg/bottle Approval method: TBD Q3W intravenous infusion (IV) sintilimab Specifications: 100mg (10ml)/bottle Afghan way: 200 mg Q3W IV infusion

SUMMARY:
The goal of this clinical trial] is toevaluate the safety, tolerability and efficacy of IBI343 combined with sintilimab in the treatment of subjects with advanced gastric/gastroesophageal junction adenocarcinoma. The main aim is to evaluate the efficacy and safety of IBI343 combination treatment in subjects with advanced gastric/gastroesophageal junction adenocarcinoma.The secondary aim is to evaluate other efficacy endpoints in subjects with IBI343 combination therapy for advanced gastric/gastroesophageal junction adenocarcinoma.The exploratory purpose is to evaluate the correlation between CLDN18.2 expression levels in tumor tissues and the efficacy of IBI343 combination therapy.

Participants will be asked to enroll about 3-12 patients in the safety introduction period.，and about 25 patients are planned to be enrolled in the POC phase.

DETAILED DESCRIPTION:
The goal of this clinical trial] is toevaluate the safety, tolerability and efficacy of IBI343 combined with sintilimab in the treatment of subjects with advanced gastric/gastroesophageal junction adenocarcinoma. The main aim is to evaluate the efficacy and safety of IBI343 combination treatment in subjects with advanced gastric/gastroesophageal junction adenocarcinoma.The secondary aim is to evaluate other efficacy endpoints in subjects with IBI343 combination therapy for advanced gastric/gastroesophageal junction adenocarcinoma.

Participants will be asked to enroll about 3-12 patients in the safety introduction period.，and about 25 patients are planned to be enrolled in the POC phase.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the written informed consent form (ICF) and be willing and able to comply with the visits and related procedures stipulated in the plan.
2. Histopathologically confirmed unresectable locally advanced, recurrent or metastatic G/GEJ AC.
3. Part 1: Previously received first-line platinum + fluorouracil + taxane systemic treatment failure or intolerance; Part 2: Previous first-line systemic standard treatment failure or intolerance.
4. According to the Response Evaluation Criteria for Solid Tumors RECIST v1.1, there is at least 1 measurable lesion (no previous radiotherapy). (Accurate measurement at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) (intravenous contrast agent is preferred) shows that its long diameter is ≥10 mm (except for lymph nodes, the short axis of the lymph node must be ≥ 15 mm), the target lesion diameter is ≥2 times the imaging slice thickness and the lesion is suitable for repeated and accurate measurement. If a lesion located in a previously irradiated area clearly demonstrates progression that meets the RECIST V1.1 criteria, the lesion can be regarded as a measurable lesion) .
5. Age ≥18 years old, no gender limit.
6. According to the Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
7. Expected survival ≥12 weeks.
8. Have adequate bone marrow and organ function:

   1. Blood routine: ANC ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L; hemoglobin content ≥ 9.0 g/dL. Subjects must not have received blood products (including red suspension) within 7 days before collecting blood samples. , platelet apheresis, cryoprecipitate, etc.), erythropoietin (EPO), G-colony stimulating factor (Granulocyte-Colony Stimulating Factor, G-CSF) or granulocyte-macrophage colony-stimulating factor (Granulocyte-Macrophage Colony-Stimulating Factor, GM-CSF) treatment;
   2. Liver function: TBIL≤1.5×ULN (TBIL≤3×ULN is allowed for subjects with Gilbert syndrome); ALT and AST for subjects without liver metastasis ≤2.5×ULN, ALT and AST for subjects with liver metastasis ≤5×ULN; albumin ≥28 g/L;
   3. Renal function: creatinine clearance ≥60 mL/min (using Cockcroft-Gault formula); urinary protein <2+ or 24h total urinary protein <1 g;
   4. Coagulation function: International Normalized Ratio (INR) ≤ 1.5 and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN (anticoagulant therapy is allowed and the coagulation function is within the above range) subjects).
9. Female subjects of childbearing age or male subjects whose partners are women of childbearing age must take effective contraceptive measures during the entire treatment period and within 6 months after the treatment period.
10. The pathological tissue test confirmed that *CLDN18.2 was positive.
11. CPS≥1.

Exclusion Criteria:

1. Are participating in another interventional clinical study, excluding observational (non-interventional) clinical studies or in the survival follow-up phase of an interventional study.
2. Receive treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor within 2 weeks or 5 half-lives (whichever is longer) before the first dose of the study drug.
3. Receive the last anti-tumor treatment 4 weeks before the first administration of the study drug or within 5 half-lives of the anti-tumor treatment drug (whichever is shorter).
4. Received therapeutic or palliative radiotherapy within 2 weeks before the first administration of the study drug.
5. Receive biliary stent implantation within 7 days before taking the study drug for the first time.
6. Plan to receive other anti-tumor treatments during the period of drug treatment in this study [Palliative radiotherapy is allowed for the purpose of relieving symptoms (such as pain) and does not affect the evaluation of efficacy].
7. Any live vaccine within 4 weeks before the first dose of study drug or planned during the study.
8. Have undergone major surgical surgery (craniotomy, thoracotomy or laparotomy or other defined by the investigator, excluding needle biopsy) or have unhealed wounds, ulcers or fractures within 4 weeks before the first administration of the study drug ; or plan to have major surgery during the study period. For palliative purposes, local surgical treatment of isolated lesions is acceptable.
9. There are toxicities caused by previous treatment that have not recovered to NCI CTCAE v5.0 grade 0 or 1 before the first administration of the study drug (excluding alopecia, fatigue, pigmentation and other toxicities that are not considered to be safety risks according to the investigator's judgment) Condition).
10. Have a history of gastrointestinal perforation and/or fistula within 6 months before the first administration of the study drug, which has not been cured after surgical treatment.
11. Presence of pyloric obstruction and/or persistent and repeated vomiting (vomiting ≥ 3 times within 24 hours).
12. Digestive tract [refers to the muscular tube from the mouth to the anal canal, including the oral cavity, pharynx, esophagus, stomach, small intestine (duodenum, jejunum, ileum), large intestine (cecum, appendix, colon, rectum) and anal canal etc.] or after endotracheal stent implantation.
13. Symptomatic central nervous system metastases. Subjects with asymptomatic brain metastases (i.e., no neurological symptoms, no need for glucocorticoid treatment, and brain metastases ≤1.5 cm) or subjects with stable symptoms after treatment of brain metastases need to meet all the following criteria to participate This study: No midbrain, pontine, cerebellar, meningeal, medulla or spinal cord metastases; clinical status remains stable for at least 4 weeks, clinical evidence confirms no new or expanding brain metastases, and corticosteroids are discontinued before the first dose of study drug and anticonvulsant medication for at least 2 weeks. Note: The central nervous system is not a target lesion.
14. Bone metastasis with risk of paraplegia.
15. Interstitial lung disease that requires steroid treatment, or a history of interstitial lung disease, non-infectious pneumonia, severely impaired lung function or uncontrolled lung disease, such as pulmonary fibrosis, severe radiation pneumonitis, acute lung disease Injury, etc., or suspected to have the above diseases during screening.
16. There are uncontrolled diseases, such as:

    1. There is an infection that is poorly controlled and requires treatment with systemic anti-infective drugs (antibiotics, antiviral drugs or antifungal drugs) within one week before the first administration of the study drug.
    2. People infected with human immunodeficiency virus (HIV) (HIV 1/2 antibody positive).
    3. Acute or chronic active hepatitis B (defined as hepatitis B surface Antigen (HBsAg) and/or hepatitis B core antibody (Hepatitis B Core Antibody, HBcAb) positive and hepatitis B virus DNA copies Number ≥ 104 copies/mL or ≥ 2000 IU/mL or acute or chronic active hepatitis C [Hepatitis C Virus antibody (HCVAb) positive, HCV RNA > 103 copies/mL]. After nucleotide antiviral treatment, low Subjects who meet the above criteria, as well as HCV antibody-positive but RNA-negative subjects are allowed to enroll.
    4. Active COVID-19 infection.
    5. Active pulmonary tuberculosis, currently receiving anti-tuberculosis treatment or receiving anti-tuberculosis treatment within 1 year before the first administration of the study drug.
    6. Active syphilis or latent syphilis requires treatment.
    7. Individuals with symptomatic congestive heart failure (New York Heart Association Class II~IV), symptomatic or poorly controlled arrhythmias, QTc interval >480 ms or congenital long/short QT syndrome or Family history.
    8. Standardize treatment for poorly controlled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg).
    9. The tumor invades or compresses surrounding important structures (such as large blood vessels, trachea, etc.) or there is a risk of gastrointestinal/respiratory fistula.
    10. Pleural effusion, ascites, or pericardial effusion that is symptomatic and requires intervention (eg, drainage).
    11. Esophageal or gastric varices requiring immediate intervention (e.g., banding or sclerotherapy) or deemed to be at higher risk for bleeding based on the opinion of the investigator or in consultation with a gastroenterologist or hepatologist, with evidence of portal hypertension (including Subjects with splenomegaly on imaging studies) or a previous history of variceal bleeding must undergo endoscopic evaluation within 3 months before the first dose of study drug.
    12. Any life-threatening bleeding event or grade 3 or 4 gastrointestinal/variceal bleeding event requiring transfusion, endoscopic or surgical treatment within 3 months before the first dose of study drug.
    13. Any arterial thromboembolic events within 6 months before the first administration of the study drug, including myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, etc.
    14. History of new or uncontrolled deep vein thrombosis, pulmonary embolism, or any other severe venous thromboembolism (implantable venous port or catheter-derived thrombosis, or Superficial venous thrombosis is not considered a "severe" venous thromboembolism).
    15. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B or more severe cirrhosis.
    16. Risk of intestinal obstruction or intestinal perforation (including but not limited to acute diverticulitis, history of abdominal abscess) or history of the following diseases: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, etc.
    17. Significant malnutrition (if intravenous nutritional supplement is required, the weight has dropped by 5% within 1 month since the signing of the informed consent form, or the weight has dropped by more than 15% within 3 months, or the food intake has been reduced by 1/2 or more within 1 week) . Exceptions will be made if malnutrition has been corrected for more than 4 weeks before the first administration of the study drug.
    18. Other acute or chronic conditions or laboratory abnormalities that may increase the risks associated with study participation or administration of study drugs, or interfere with the interpretation of study results, and which, in the investigator's discretion, would result in the subject being classified as Not eligible to participate in this study.
    19. Neurological, psychiatric or social conditions that affect compliance with study requirements, significantly increase the risk of AEs, or affect the subject's ability to provide written ICF.
17. History of other primary malignant tumors, except for the following:

    * Cured malignancy, no known active disease for ≥2 years before study enrollment and extremely low risk of recurrence;
    * Nonmelanoma skin cancer or lentigo maligna that has been adequately treated and without evidence of disease recurrence;
    * Carcinoma in situ that has been adequately treated and without evidence of disease recurrence.
18. Known history of immunodeficiency.
19. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
20. Long-term use of systemic hormones or immunosuppressive drugs that are not reduced to physiological doses or discontinued 4 weeks before the first dose, excluding: intranasal inhaled local steroid treatment or local steroid injection (such as intra-articular injection) ; Systemic corticosteroid treatment not exceeding 10 mg/day of prednisone or its equivalent physiological dose; Glucocorticoids as preventive medication for allergic reactions (such as medication before CT) and vomiting prevention medication specified in the protocol. Requires long-term systemic corticosteroids or any other immunosuppressive drug therapy, excluding inhaled corticosteroids.
21. Suffering from active autoimmune diseases or inflammatory diseases [including inflammatory bowel disease (such as ulcerative colitis, Crohn's disease, etc.), celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome or Wegener syndrome ( Granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.], or a history of this disease within the past 2 years. Subjects with vitiligo, psoriasis, alopecia or Grave's disease who do not require systemic treatment within the past 2 years, hypothyroidism who only require thyroid hormone replacement therapy, and type 1 diabetes who only require insulin replacement therapy can be enrolled. . Subjects who are only positive for autoimmune antibodies need to confirm whether there is an autoimmune disease according to the researcher's judgment.
22. Previous treatment with antibody drug conjugates based on topoisomerase inhibitors.
23. For subjects receiving drug treatment, there is a history of allergy to corresponding drugs or preparations.
24. For subjects receiving drug treatment, there are contraindications to the corresponding drugs.
25. For subjects receiving drug treatment, there has been a history of adverse reactions related to the corresponding drugs that led to permanent discontinuation of the drug.
26. Pregnant or lactating female subjects.
27. Other researchers believe that you are not eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  Objective Response Rate (ORR) evaluated according to RECIST v1.1.
AE | 24 months
  Adverse Event (AE), changes and incidence rates and their correlation with experimental drugs.
Treatment-Emergent Adverse Event (TEAE) | 24 months
  Treatment-Emergent Adverse Event (TEAE) changes and incidence rates and their correlation with experimental drugs.
Adverse Event of Special Interest (AESI) | 24 months
  Adverse Event of Special Interest (AESI) changes and incidence rates and their correlation with experimental drugs.
Serious Adverse Event (SAE) | 24 months
  Serious Adverse Event (SAE) changes and incidence rates and their correlation with experimental drugs.
laboratory examinations | 24 months
  laboratory examinations changes and incidence rates and their correlation with experimental drugs.
physical examinations | 24 months
  physical examinations changes and incidence rates and their correlation with experimental drugs.
vital signs | 24 months
  vital signs, etc.changes and incidence rates and their correlation with experimental drugs.

SECONDARY OUTCOMES:
PFS | 24 months
  Progression-free Survival (PFS)
Duration of Response (DoR) | 24 months
  Duration of Response (DoR)
Disease Control Rate (DCR) | 24 months
  Disease Control Rate (DCR)
Time to Response (TTR) | 24 months
  Time to Response (TTR)
Overall Survival (OS) | 24 months
  Overall Survival (OS)

OTHER OUTCOMES:
CLDN18.2 expression level | 24 months
  CLDN18.2 expression level in tumor tissue at baseline and its relationship with efficacy.

IPD SHARING:
Plan to Share IPD: No